CLINICAL TRIAL: NCT04644393
Title: Responsiveness and Validation Study of MFM-20 in SMA Patients Treated With Nusinersen: Retro NusiMFM
Brief Title: Responsiveness and Validation Study of MFM-20 in SMA Patients Treated With Nusinersen
Acronym: RetroNusiMFM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_1086
Record Dates: First submitted 2020-11-20; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; Motor Function Measure; Outcome Assessment; Nusinersen
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Motor Function Measure (MFM), a reliable tool assessing motor function and its progression in most neuromuscular diseases, is widely used in France in many teams. It can be used regardless of the severity of the motor impairment or the ambulatory status of the patient, allowing its use throughout the whole follow-up period of the patient, even in case of the loss of walking. Two versions of the MFM exist, one composed of 32 items validated for patients from 6 years old (MFM-32) and a shorter version composed of 20 items validated for patients between 2 and 6 years old (MFM-20).

In order to show the possible use of MFM-20 as early as the age of 2 years to validly and reliably monitor the evolution of the motor function of children treated with Nusinersen, we propose in this project to study the sensitivity to treatment-induced change of MFM-20 and the validity of the scale in this population.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls with Type 1 or 2 Spinal Muscular Atrophy, genetically confirmed
* Aged 2 to 6 years old
* Treated by Nusinersen for at least two months
* With at least 3 MFM-20 repeated measures, and with adelay minimum between the first and the last MFM-20 of 6 months
* With parental assent

Exclusion Criteria:

* - Patients with associated cognitive impairment making impossible evaluation of motor function
* Patients participating to a clinical study with a potential effect on their motor function.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: * Boys and girls with Type 1 or 2 Spinal Muscular Atrophy, genetically confirmed
  * Aged 2 to 6 years old
  * Treated by Nusinersen for at least two months
  * With at least 3 MFM-20 repeated measures, and with adelay minimum between the first and the last MFM-20 of 6 months
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
MFM-20 responsiveness | At least 6 Months after the first MFM-20 assessment, and at maximum 24 months
  The MFM-20 sensitivity to change indexes considered will be the effect amplitude and the Standardized Response Mean (SRM).

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Service de neuropédiatrie et neurochirurgie de l'enfant Centre de Référence maladies neuromusculaires AOC CHU d'Angers, Angers
  - Service de génétique médicale Pôle de Pédiatrie CHU Estaing, Clermont-Ferrand
  - Service de Neurologie et réanimation pédiatriques CHU Paris IdF Ouest - Hôpital Raymond Poincaré, Garche
  - Hospices Civils de Lyon, Hôpital Femme Mère Enfant, Lyon
  - Apf Esean, Nantes
  - Institut I-Motion - Centre de recherche pédiatrique en pathologies neuromusculaires CHU Paris Est - Hôpital d'Enfants Armand-Trousseau, Paris
  - Service de pédiatrie CHU de Saint-Etienne, Saint-Priest-en-Jarez
  - Unité de Neurologie Pédiatrique Centre de Référence Maladies NeuroMusculaires Hôpital des Enfants CHU Toulouse, Toulouse